CLINICAL TRIAL: NCT04786106
Title: Comparison of Collagenase Clostridium Histolyticum to Surgery for the Management of Peyronie's Disease: A Randomized Trial
Brief Title: Investigation of Surgery, Collagenase, and Restorex for the Improvement of Peyronie's
Acronym: iSCRIP
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Charitable Union for the Research and Education of Peyronie's Disease (Other)
Collaborators: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CUREPD101
Record Dates: First submitted 2021-02-05; First posted 2021-03-08 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Peyronie's Disease
Keywords: collagenase clostridium histolyticum; RestoreX; plication; incision and grafting; surgery
MeSH Terms: conditions — Penile Induration; Surgical Wound | interventions — Microbial Collagenase; Transplantation; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The curvature and length assessments will be performed without knowledge as to pre-treatment measurements.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CCH+PTT (Active Comparator): Men will receive two injections of CCH administered 1-3 days apart, followed by manual modeling and PTT 30-60 min/day as outlined in our prior publication. Approximately 6 weeks later, the next round of injections will be performed until a maximum of 8 injections in total has been administered. PTT will be continued until the 3-month post-treatment visit.
  Interventions: Drug: Collagenase Clostridium Histolyticum 0.9 MG [Xiaflex] (CCH); Device: RestoreX Penile Traction Device
- Surgery+PTT (Active Comparator): Men will undergo either penile plication or I&G based on appropriate clinical criteria for either surgery. 2-4 weeks post-operatively (depending on tolerability), the patients will be asked to perform PTT 30-60 minutes daily until the 3-month post-treatment visit.
  Interventions: Procedure: Penile Plication Surgery; Procedure: Incision and Grafting (I&G) Surgery; Device: RestoreX Penile Traction Device

INTERVENTIONS:
Drug: Collagenase Clostridium Histolyticum 0.9 MG [Xiaflex] (CCH) — Men in this cohort would receive the full series of 8 Xiaflex injections: 2 injections separated by 1-3 days, repeated 3 additional times with 6 week breaks between treatments.
  Other Names: Xiaflex
  Arms: CCH+PTT
Procedure: Penile Plication Surgery — Men in this cohort would undergo surgery using either penile plication or incision and grafting. The specific surgery would be selected based on commonly used criteria: plication for curvatures <70 degrees; I&G used for ≥70 degrees or severe hourglass / hinge deformities. However, the specific surgery (plication vs I&G) will ultimately be decided based on the primary investigator's clinical judgment.
  Arms: Surgery+PTT
Procedure: Incision and Grafting (I&G) Surgery — Men in this cohort would undergo surgery using either penile plication or incision and grafting. The specific surgery would be selected based on commonly used criteria: plication for curvatures <70 degrees; I&G used for ≥70 degrees or severe hourglass / hinge deformities. However, the specific surgery (plication vs I&G) will ultimately be decided based on the primary investigator's clinical judgment.
  Arms: Surgery+PTT
Device: RestoreX Penile Traction Device — RestoreX is a Class I PTT device developed by PathRight Medical, is registered with the FDA, and has randomized controlled data demonstrating efficacy when used for the treatment of PD.

SUMMARY:
The purpose of this study is to compare key clinical outcomes of collagenase clostridium histolyticum injections versus surgery for the management of Peyronie's Disease.

DETAILED DESCRIPTION:
After eligible patients have been informed about the study protocol and risks and consent have been given, men will be randomly assigned into either the collagenase clostridium histolyticum + penile traction therapy (CCH + PTT) group or to the surgery + penile traction therapy (surgery + PTT) group. Those in the CCH + PTT group will receive the full 4 series of 8 Xiaflex injections with 1-3 days between each set of 2 injections and 6 weeks prior to the next series. Patients would then use the RestoreX traction device throughout the series to 3 months post-treatment. Those that were assigned the surgery + PTT treatment protocol would undergo surgery using either penile plication or incision and grafting, depending on the degree of curvature and erectile function. Traction using RestoreX will also be prescribed to these men 2-4 weeks post-operatively until 3 months post-treatment. Key clinical outcomes of both treatment protocols will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Men with PD
* >18 years old
* Curvature ≥30 degrees
* Ability to achieve an erection satisfactory for intercourse with or without PDE5 inhibitors

Exclusion Criteria:

* Prior treatment with CCH or surgery
* Moderate (shadowing) or severe (>1 cm) penile calcification
* Any contraindications to CCH, PTT, or surgery - as determined by the PI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-30 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Overall satisfaction with treatment | 1 year
  Answer to SAPS question #1 (How satisfied are you with the effect of your treatment?) to determine overall satisfaction at all time points
Subjective reporting of erectile dysfunction post treatment | 1 year
  Comparison of erectile dysfunction complication rates
Subjective reporting of changes in penile sensation post treatment | 1 year
  Comparison of changes in penile sensation complication rates
Subjective reporting of changes in penile length post treatment | 1 year
  Comparison of perceived changes in penile length complication rates
International Index of Erectile Function, Erectile Function Domain (IIEF) Scores | 1 year
  Comparison of IIEF erectile function domain score (Q1-5, 15; min/max 1-30; higher is better)

SECONDARY OUTCOMES:
Peyronie's Disease Questionnaire (PDQ) Scores | 1 year
  Comparison of PDQ questionnaire scores; Subdomains - psychological and physical (Q1-6; min/max 0-24; lower is better), penile pain (Q7-9; min/max 0-30; lower is better), symptom bother (Q10-15; min/max 0-16; lower is better)
International Index of Erectile Function (IIEF) Scores | 1 year
  Comparison of IIEF questionnaire scores-all domains except erectile function (which is a primary endpoint); subdomains: orgasmic function (Q9-10; min/max 0-10; higher is better), sexual desire (Q11-12; min/max 2-10; higher is better), intercourse satisfaction (Q6-8; min/max 0-15; higher is better), overall satisfaction (Q13-14; min/max 2-10; higher is better)
Beck's Depression Inventory (BDI) Scores | 1 year
  Comparison of BDI questionnaire scores on depression. 21 items (min/max 0-63, lower is better)
Penile Curvature | 1 year
  Comparison of changes in penile curvature
Objective measurements of penile length post treatment (compared to pre-treatment) | 1 year
  Comparison of changes in penile length
Interventions required | 1 year
  Comparison of subsequent interventions required - surgery or CCH injections
Hospitalizations | 1 year
  Number of hospitalizations or ER visits resulting from treatment
Non-standardized questionnaire | 1 year
  Comparison of non-standardized questionnaire responses

CONTACTS AND LOCATIONS:
Locations (1):
- The Male Fertility and Peyronie's Clinic, Orem, Utah, United States

DOCUMENTS (2):
  • Study Protocol (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/06/NCT04786106/Prot_000.pdf
  • Informed Consent Form (2020-12-28): https://cdn.clinicaltrials.gov/large-docs/06/NCT04786106/ICF_001.pdf